CLINICAL TRIAL: NCT03112512
Title: A Comparison of Optimal Positive End-expiratory Pressure Determination Guided by Electrical Impedance Tomography and Protective Ventilation Tool by G5(MV) in Moderate and Severe Acute Respiratory Distress Syndrome Patients
Brief Title: A Comparison of Optimal PEEP Determination Guided by EIT and G5 Device in Moderate and Severe ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mei-Yun Chang (Other)
Responsible Party: Sponsor-Investigator, Mei-Yun Chang, Principal Investigator, Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FEMH-105117-E
Record Dates: First submitted 2017-03-15; First posted 2017-04-13 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: optimal positive end-expiratory pressure determination; Electrical impedance tomography
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT (Experimental): PEEP titration is performed where EIT is measured at the same time. After PEEP titration, EIT data is analyzed. Global inhomogeneity index and regional compliance based on EIT are calculated. PEEP level is selected when ventilation distribution is most homogeneous.
  Interventions: Device: optimal PEEP guided by EIT
- G5 VENTILATOR (Experimental): Protective Ventilation Tool by G5(MV) to determine the optimal PEEP on ARDS patients. The results are delivered by the ventilator automatically.
  Interventions: Device: optimal PEEP guided by G5 ventilator

INTERVENTIONS:
Device: optimal PEEP guided by EIT — Patients are randomly assigned to EIT group or G5 group. PEEP selected in EIT group is based on GI index and regional compliance. PEEP decided in G5 group is based on the ventilator.
  Arms: EIT
Device: optimal PEEP guided by G5 ventilator — Patients are randomly assigned to EIT group or G5 group. PEEP selected in EIT group is based on GI index and regional compliance. PEEP decided in G5 group is based on the ventilator.
  Arms: G5 VENTILATOR

SUMMARY:
To Select the Optimal Positive End-expiratory Pressure in Moderate and Severe Acute Respiratory Distress Syndrome Patients by Using:

1. the novel Non-invasive Electrical Impedance Tomography Guided Method
2. the Protective ventilation tool G5(MV)

DETAILED DESCRIPTION:
1. To titrate PEEP guided by EIT. A global inhomogeneity (GI) index and regional compliance based on EIT were developed to quantify the tidal volume distribution within the lung. The aim of this study was to test the feasibility of optimizing PEEP with respect to ventilation homogeneity using the GI index and regional compliance.
2. To titrate PEEP with the Protective Ventilation Tool by G5(MV). The new generation of ventilator will deliver an optimal PEEP on ARDS patients based on their status automatically.

ELIGIBILITY:
Inclusion Criteria:

1. ARDS patients
2. Transferred from FEMH emergency room or Ward into the medical intensive care unit.
3. Patients with invasive mechanical ventilation
4. Patient, agent or consent of families learn about and subjects were willing to sign the consent form.

Exclusion Criteria:

1. burning electric knife used
2. pacemaker used
3. Large area wound is used gauze to cover
4. Wound or burn injuries of the chest wall.
5. Patients included conditions are not met.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 20-90 years old
Enrollment: 88 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Respiratory system parameter | 48 hrs
  Compliance

SECONDARY OUTCOMES:
MV day | 64 days
  Number of days with ventilator and ICU stay
Respiratory system parameter | 48 hrs
  PaO2/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Chang MEI YUN, MASTER, Principal Investigator — FEMH -chest division
Locations (1):
- Electrical impedance tomography (EIT), New Taipei City, No.21, Sec. 2, Nanya S. Rd., Banciao Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No
no sharing plan, including what IPD are to be shared with other researchers

REFERENCES:
- [Result] Franchineau G, Brechot N, Lebreton G, Hekimian G, Nieszkowska A, Trouillet JL, Leprince P, Chastre J, Luyt CE, Combes A, Schmidt M. Bedside Contribution of Electrical Impedance Tomography to Setting Positive End-Expiratory Pressure for Extracorporeal Membrane Oxygenation-treated Patients with Severe Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2017 Aug 15;196(4):447-457. doi: 10.1164/rccm.201605-1055OC. PMID 28103448
- [Derived] Hsu HJ, Chang HT, Zhao Z, Wang PH, Zhang JH, Chen YS, Frerichs I, Moller K, Fu F, Hsu HS, Chuang SP, Hsia HY, Yen DH. Positive end-expiratory pressure titration with electrical impedance tomography and pressure-volume curve: a randomized trial in moderate to severe ARDS. Physiol Meas. 2021 Feb 6;42(1):014002. doi: 10.1088/1361-6579/abd679. PMID 33361553
- [Derived] Zhao Z, Lee LC, Chang MY, Frerichs I, Chang HT, Gow CH, Hsu YL, Moller K. The incidence and interpretation of large differences in EIT-based measures for PEEP titration in ARDS patients. J Clin Monit Comput. 2020 Oct;34(5):1005-1013. doi: 10.1007/s10877-019-00396-8. Epub 2019 Oct 5. PMID 31587120
- [Derived] Zhao Z, Chang MY, Chang MY, Gow CH, Zhang JH, Hsu YL, Frerichs I, Chang HT, Moller K. Positive end-expiratory pressure titration with electrical impedance tomography and pressure-volume curve in severe acute respiratory distress syndrome. Ann Intensive Care. 2019 Jan 17;9(1):7. doi: 10.1186/s13613-019-0484-0. PMID 30656479
- See also: Bedside Contribution of Electrical Impedance Tomography to Set Positive End-Expiratory Pressure for ECMO-Treated Severe ARDS Patients. — https://www.ncbi.nlm.nih.gov/pubmed/28103448